CLINICAL TRIAL: NCT01693588
Title: The Effect of a Multimodality Pain Management Protocol on Postoperative Neurosurgical Pain
Brief Title: Study of a Multimodality Pain Management Protocol on Postoperative Neurosurgical Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 341-2012
Record Dates: First submitted 2012-09-14; First posted 2012-09-26 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Pain; Postoperative Pain; Surgical Pain; Neurosurgical Pain
Keywords: Pain; Postoperative Pain; Surgical Pain; Neurosurgical Pain
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pain Management Bundle (Experimental): The Pain Management Bundle will be implemented for all postoperative neurosurgical patients admitted to nursing units at the University of Florida.
  Interventions: Other: Pain Management Bundle

INTERVENTIONS:
Other: Pain Management Bundle — The Pain Management Bundle will be implemented for all postoperative neurosurgical patients admitted to nursing units at the University of Florida.

SUMMARY:
High levels of postoperative pain are associated with an increased risk of lung and heart complications, are the most common reason for delayed discharge or for unexpected hospital admission after ambulatory surgery, and are responsible for prolonged recovery after inpatient surgery. Furthermore both neuropathic pain and post surgical pain inhibit weight gain and may have an impact on the patient's nutrition post operatively. The purpose of this study is to evaluate the effectiveness of a multimodality pain management protocol on postoperative neurosurgical pain.

DETAILED DESCRIPTION:
Despite the long-standing recognition of postoperative pain as both prevalent and undertreated, 20% to 30% of all surgical patients continue to experience moderate to severe postoperative pain. High levels of postoperative pain are associated with an increased risk of pulmonary and cardiovascular complications, are the most common reason for delayed discharge or for unexpected hospital admission after ambulatory surgery, and are responsible for prolonged convalescence after inpatient surgery. Furthermore both neuropathic pain and post surgical pain inhibit weight gain and may have an impact on the patient's nutrition post operatively. Finally, high levels of postoperative pain have also been associated with an increased risk of chronic pain. Therefore, the aggressive treatment of postoperative pain may be particularly important in influencing patient outcomes, inadvertent readmissions, and propensity for developing chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Postoperative neurosurgical patient treated at the University of Florida
* Primary language is English

Exclusion Criteria:

* Younger than 18 or older than 100 years of age
* Patients who are pregnant, wards of the state, prisoners, and patients who lack the ability to communicate their pain level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Mean Score on the Visual Analogue Scale | Post Operative Day 1
  The Visual Analogue Scale measures the severity of pain on a continuous scale from 0 (no pain) to 10 (worst possible pain).
Mean Score on the Visual Analogue Scale | Post Operative Day 3
  The Visual Analogue Scale measures the severity of pain on a continuous scale from 0 (no pain) to 10 (worst possible pain).

SECONDARY OUTCOMES:
Score on the HCAHP survey. | Hospital discharge, an expected average of 5 days.
  The HCAHP survey measures how often patients perceived an aspect of their care was performed, generally using a scale of always, usually, sometimes, and never.

CONTACTS AND LOCATIONS:
Overall Officials: William L. Titsworth, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Titsworth WL, Abram J, Guin P, Herman MA, West J, Davis NW, Bushwitz J, Hurley RW, Seubert CN. A prospective time-series quality improvement trial of a standardized analgesia protocol to reduce postoperative pain among neurosurgery patients. J Neurosurg. 2016 Dec;125(6):1523-1532. doi: 10.3171/2015.10.JNS15698. Epub 2016 Mar 11. PMID 26967774